CLINICAL TRIAL: NCT00081562
Title: Family Studies of the Genetics of Ankylosing Spondylitis
Brief Title: Genetics of Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Other Study IDs: NIAMS-098; 5R01AR046208-05 (NIH); NASC
Record Dates: First submitted 2004-04-15; First posted 2004-04-19 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Spondylitis; Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis; Spondylitis, Ankylosing

SUMMARY:
Ankylosing spondylitis (AS) is a chronic inflammatory disease that affects the joints between the vertebrae of the spine and the joints between the spine and the pelvis. The purpose of this study is to collect information and blood samples from patients with AS and their relatives for use in genetic studies.

DETAILED DESCRIPTION:
AS is a chronic inflammatory disease that eventually causes the affected vertebrae to fuse or grow together. The cause of AS is unknown, but genetic factors seem to play a role. Risk factors include a family history of ankylosing spondylitis and male gender.

This study will collect patient information and blood samples from affected patients (and when available, both parents of the affected patients) of 400 families with children fulfillling the modified New York criteria for AS. Diagnosis of AS will be verified by patient questionnaire, medical record review, and pelvic radiographs. Information from these patients will be used to search the human genome for disease-associated loci and/or genes. This study will also utilize contributions of investigators who have conducted recent clinical or genetic research in AS at 10 academic medical centers throughout North America (the North American Spondylitis Consortium, or NASC).

ELIGIBILITY:
Inclusion Criteria:

* Meet modified New York criteria for ankylosing spondylitis (AS)
* AS as confirmed by X-rays of sacroiliac joints (between the pelvis and spine)
* At least two siblings in family with AS
* Parents of the participants with AS have the option of also being enrolled

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600
Dates: Start 1999-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Reveille, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Texas - Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Background] Brown MA, Wordsworth BP, Reveille JD. Genetics of ankylosing spondylitis. Clin Exp Rheumatol. 2002 Nov-Dec;20(6 Suppl 28):S43-9. PMID 12463446
- [Background] Tsui FW, Tsui HW, Cheng EY, Stone M, Payne U, Reveille JD, Shulman MJ, Paterson AD, Inman RD. Novel genetic markers in the 5'-flanking region of ANKH are associated with ankylosing spondylitis. Arthritis Rheum. 2003 Mar;48(3):791-7. doi: 10.1002/art.10844. PMID 12632434
- [Background] Reveille JD. The genetic basis of spondyloarthritis. Curr Rheumatol Rep. 2004 Apr;6(2):117-25. doi: 10.1007/s11926-004-0056-6. PMID 15016342
- See also: Click here for the North American Spondylitis Consortium [NASC] Web site. — http://www.asresearch.org
- See also: Click here for the Spondylitis Association of America Web site. — http://www.spondylitis.org/